CLINICAL TRIAL: NCT02913482
Title: A Two Part Seamless, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Risdiplam (RO7034067) in Infants With Type 1 Spinal Muscular Atrophy
Brief Title: Investigate Safety, Tolerability, PK, PD and Efficacy of Risdiplam (RO7034067) in Infants With Type1 Spinal Muscular Atrophy
Acronym: FIREFISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP39056; 2016-000778-40 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Finding): Risdiplam (RO7034067) (Experimental): Participants will receive multiple ascending doses of risdiplam (RO7034067), administered orally once daily for a minimum of 4 weeks to select the dose for Part 2. During the first year of treatment, most participants will switch to the Part 2 dose. During the second year of treatment, all Part 1 participants will be receiving the Part 2 dose. They will thereafter enter a 3-year open-label extension phase and continue to receive risdiplam at the same dose.
  Interventions: Drug: Risdiplam
- Part 2 (Confirmatory): Risdiplam (RO7034067) (Experimental): Participants will receive risdiplam (RO7034067), administered orally once daily at the dose defined in Part 1 of the study, for a duration of 24 months. They will thereafter enter a 3-year open-label extension phase and continue to receive risdiplam at the same dose.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Risdiplam will be administered orally.
  Other Names: RO7034067, Evrysdi

SUMMARY:
Open-label, multi-center clinical study is to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamics (PD), and efficacy of Risdiplam (RO7034067) in infants with Type 1 spinal muscular atrophy (SMA). The study consists of two parts, an exploratory dose finding part (Part 1) and a confirmatory part (Part 2) which will investigate Risdiplam (RO7034067) for 24-months at the dose selected in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history, signs or symptoms attributable to Type 1 SMA with onset after 28 days but prior to the age of 3 months
* Gestational age of 37 to 42 weeks
* Confirmed diagnosis of 5q-autosomal recessive SMA
* Participants has two survival motor neuron 2 (SMN2) gene copies, as confirmed by central testing
* Body weight greater than or equal to (>=) third percentile for age, using appropriate country-specific guidelines
* Receiving adequate nutrition and hydration (with or without gastrostomy) at the time of screening, in the opinion of the Investigator
* Adequately recovered from any acute illness at the time of screening and considered well-enough to participate in the opinion of the Investigator

Exclusion Criteria:

* Concomitant or previous participation in any investigational drug or device study within 90 days prior to screening or 5 half-lives, whichever is longer
* Concomitant or previous administration of SMN2-targeting antisense oligonucleotide, SMN2 splicing modifier or gene therapy study
* Any history of cell therapy
* Hospitalization for pulmonary event within the last 2 months, or planned at the time of screening
* Presence of clinically relevant electrocardiogram (ECG) abnormalities before study drug administration
* Unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system diseases
* Participants requiring invasive ventilation or tracheostomy
* Participants requiring awake non-invasive ventilation or with awake hypoxemia (arterial oxygen saturation less than [<] 95 percent [%]) with or without ventilator support
* Participants with a history of respiratory failure or severe pneumonia, and have not fully recovered their pulmonary function at the time of screening
* Multiple or fixed contractures and/or hip subluxation or dislocation at birth
* Presence of non-SMA related concurrent syndromes or diseases
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first dose administration
* Any inhibitor of cytochrome P450 (CYP) 3A4 and/or any Organic Cation Transporter 2 (OCT-2) and multidrug and toxin extrusion (MATE) substrates taken within 2 weeks and/or any inducer of CYP3A4 taken within 4 weeks (or within 5-times the elimination half-life, whichever is longer) prior to dosing or participants (and the mother, if breastfeeding the infant) taking any nutrients known to modulate CYP3A activity and any known flavin containing monooxygenase (FMO) 1 or FMO3 inhibitors or substrates
* Prior use (at any time in the participants lives) and/or anticipated need for quinolones (chloroquine and hydroxychloroquine), thioridazine, vigabatrin, retigabine, or any other drug known to cause retinal toxicity during the study. Infants exposed to chloroquine, hydroxycholoroquine, thioridazine, vigabatrin, retigabine or drugs with known retinal toxicity given to mothers during pregnancy (and lactation) should not be enrolled.
* Recent history (less than 6 months) of ophthalmic disease that would interfere with the conduct of the study as assessed by an ophthalmologist
* Therapeutic use, defined as use for 8 weeks or longer, of the following medications within 90 days prior to enrollment: riluzole, valproic acid, hydroxyurea, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, probenecid, agents anticipated to increase or decrease muscle strength, agents with known or presumed histone deacetylase (HDAC) inhibitory effect, medications known to or suspected of causing retinal toxicity (deferoxamine, topiramate, latanoprost, niacin, rosiglitazone, tamoxifen, canthaxanthine, sildenafil, and interferon) and medications with known phototoxicity liabilities (e.g., oral retinoids including over-the-counter [OTC] formulations, amiodarone, phenothiazines and use of minocycline)

Ages: 1 Month to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (4):
  - Stanford University Medical Center, Palo Alto, California
  - Ann and Robert H. Lurie Children Hospital of Chicago, Chicago, Illinois
  - Boston Childrens Hospital, Boston, Massachusetts
  - Columbia University Medical Center; The Neurological Institute of New York, New York, New York
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
- Brazil (2):
  - Instituto de Puericultura E Pediatria Martagão Gesteira, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - FMUSP_X; Neurologia, São Paulo, São Paulo
- China (2):
  - Peking University First Hospital, Beijing
  - Children's Hospital of Fudan University, Shanghai
- Clinical Medical Center Zagreb; University Hospital Rebro Department of Paediatrics, Zagreb, Croatia
- France (2):
  - Hopital Femme Mere Enfant; Medecine Physique et Readaptation Pediatrique ? L?ESCALE, Bron
  - Hopital Armand Trousseau, Paris
- Italy (5):
  - IRCCS Ospedale Pediatrico Bambino Gesù; U.O. Malattie Neuromuscolari e Neurodegenerative, Rome, Lazio
  - Policlinico Agostino Gemelli; Dipartimento di Neuropsichiatria Infantile, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini; U.O.S.D. Centro di Miologia e Patologie Neurodegenerative, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico; Unità Operativa Complessa di Neurologia, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico ?Carlo Besta?; UO di Neurologia dello Sviluppo, Milan, Lombardy
- Hyogo Medical University Hospital, Hyōgo, Japan
- Poland (2):
  - Szpital Gdanskiego Uniwersytetu Medycznego; Clinic of developmental neurology, Gda?sk
  - The Children?s Memorial Health Institute Department of Neurology and Epileptology, Warsaw
- Russian Children Neuromuscular Center of Veltischev, Moscow, Moscow Oblast, Russia
- King Faisal Specialist Hospital and Research Centre Building, Riyadh, Saudi Arabia
- Institute for Mother and Child Dr. Vukan Cupic, Belgrade, Serbia
- Spain (3):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari Vall d'Hebron; Area Genética Clínica y Molecular, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- Universitäts-Kinderspital (UKBB) Neuropädiatrie, Basel, Switzerland
- Turkey (Türkiye) (2):
  - Hacettepe University, School of Medicine; Pediatrics Department; Pediatrics Child Neurology Unit, Ankara
  - Hospital Yeditepe University Kozyatagi; Pediatry, Atasehir- Istanbul
- Ams of Ukraine; Inst. of Neurology, Psychiatry & Narcology, Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Cleary Y, Kletzl H, Grimsey P, Heinig K, Ogungbenro K, Silber Baumann HE, Frey N, Aarons L, Galetin A, Gertz M. Estimation of FMO3 Ontogeny by Mechanistic Population Pharmacokinetic Modelling of Risdiplam and Its Impact on Drug-Drug Interactions in Children. Clin Pharmacokinet. 2023 Jun;62(6):891-904. doi: 10.1007/s40262-023-01241-7. Epub 2023 May 6. PMID 37148485
- [Derived] Masson R, Mazurkiewicz-Beldzinska M, Rose K, Servais L, Xiong H, Zanoteli E, Baranello G, Bruno C, Day JW, Deconinck N, Klein A, Mercuri E, Vlodavets D, Wang Y, Dodman A, El-Khairi M, Gorni K, Jaber B, Kletzl H, Gaki E, Fontoura P, Darras BT; FIREFISH Study Group. Safety and efficacy of risdiplam in patients with type 1 spinal muscular atrophy (FIREFISH part 2): secondary analyses from an open-label trial. Lancet Neurol. 2022 Dec;21(12):1110-1119. doi: 10.1016/S1474-4422(22)00339-8. Epub 2022 Oct 14. PMID 36244364
- [Derived] Cances C, Vlodavets D, Comi GP, Masson R, Mazurkiewicz-Beldzinska M, Saito K, Zanoteli E, Dodman A, El-Khairi M, Gorni K, Gravestock I, Hoffart J, Scalco RS, Darras BT; ANCHOVY Working Group. Natural history of Type 1 spinal muscular atrophy: a retrospective, global, multicenter study. Orphanet J Rare Dis. 2022 Jul 29;17(1):300. doi: 10.1186/s13023-022-02455-x. PMID 35906608
- [Derived] Darras BT, Masson R, Mazurkiewicz-Beldzinska M, Rose K, Xiong H, Zanoteli E, Baranello G, Bruno C, Vlodavets D, Wang Y, El-Khairi M, Gerber M, Gorni K, Khwaja O, Kletzl H, Scalco RS, Fontoura P, Servais L; FIREFISH Working Group. Risdiplam-Treated Infants with Type 1 Spinal Muscular Atrophy versus Historical Controls. N Engl J Med. 2021 Jul 29;385(5):427-435. doi: 10.1056/NEJMoa2102047. PMID 34320287
- [Derived] Baranello G, Darras BT, Day JW, Deconinck N, Klein A, Masson R, Mercuri E, Rose K, El-Khairi M, Gerber M, Gorni K, Khwaja O, Kletzl H, Scalco RS, Seabrook T, Fontoura P, Servais L; FIREFISH Working Group. Risdiplam in Type 1 Spinal Muscular Atrophy. N Engl J Med. 2021 Mar 11;384(10):915-923. doi: 10.1056/NEJMoa2009965. Epub 2021 Feb 24. PMID 33626251
- See also: roche-sma-clinicaltrials.com provides information about the Roche Firefish clinical trial NCT02913482 and molecule being investigated in SMA. — http://roche-sma-clinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 was conducted at 7 investigational sites across 5 countries; Part 2 was conducted at 14 investigational sites across 10 countries.
Groups:
- Exploratory Part 1 - Cohort 1: Participants received risdiplam in a staggered, dose-escalation manner once daily at Dose Level 1 for a minimum of 4 weeks to select the dose for Part 2. Dose Level 1 was targeting an exposure of mean AUC0-24h,ss 700 ng*h/mL.
- Exploratory Part 1 - Cohort 2: Participants received risdiplam in a staggered, dose-escalation manner once daily at Dose Level 2 for a minimum of 4 weeks to select the dose for Part 2. Dose Level 2 was targeting an exposure of mean AUC0-24h,ss </= 2000 ng*h/mL.
- Confirmatory Part 2 - Risdiplam: Participants received risdiplam orally once daily at a dose targeting an exposure of mean AUC0-24h,ss </= 2000 ng*h/mL, for a duration of 24 months with a primary analysis after 12 months. Starting doses were either 0.04mg/kg, 0.08mg/kg or 0.2mg/kg depending on the participant's age. All participants had their dose adjusted to 0.2mg/kg within a few months of starting treatment. The dose was adjusted to 5 mg when the participant reached 20 kg body weight.
Period: Overall Study
Arm/Group | Exploratory Part 1 - Cohort 1 | Exploratory Part 1 - Cohort 2 | Confirmatory Part 2 - Risdiplam
Started | 4 | 17 | 41
Completed | 3 | 13 | 36
Not Completed | 1 | 4 | 5
Not completed — Death | 0 | 2 | 2
Not completed — Progressive Disease | 1 | 1 | 1
Not completed — Reason not specified | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exploratory Part 1 - Cohort 1 | Exploratory Part 1 - Cohort 2 | Confirmatory Part 2 - Risdiplam | Total
Number analyzed (Participants) | 4 | 17 | 41 | 62
Age, Continuous [Mean (Standard Deviation); unit: Months] | 6.84 (0.10) | 5.56 (1.43) | 5.20 (1.47) | 5.41 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 22 | 37
  Male | 0 | 6 | 19 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 4 | 17 | 36 | 57
  Hispanic or Latino | 0 | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 4 | 14 | 18
  White | 4 | 9 | 22 | 35
  Unknown | 0 | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Selected Part 2 Dose of Risdiplam
Description: All safety, tolerability, PK and PD data available up to the clinical cut-off date of 5 January 2018, plus data that became available prior to the database snapshot on 6 February 2018 were included in the Internal Monitoring Committee (IMC) review. The IMC was responsible for selecting the dose for Part 2 of the study (pivotal dose). An external Independent Data Monitoring Committee (iDMC) reviewed data from Part 1 and confirmed the dose-selection decision of the IMC. The dose for Part 2 selected by the IMC was a dose that: 1.Was judged to be safe and well-tolerated, based on all available safety data from Part 1 and as confirmed by the iDMC; 2. Resulted in an exposure at steady-state below the exposure cap (mean value) of AUC0-24h,ss 2000 ng*h/mL (adjusted for free-fraction, if required); 3. Resulted in an SMN protein increase that was expected to be clinically relevant.
Time Frame: Minimum of 2 weeks at steady state exposure
Population: All participants in Part 1 who received at least one dose of risdiplam and had available data at the time of the data snapshot for selecting the Part 2 dose.
Measure: Number; unit: mg/kg
Groups:
- Exploratory Part 1 - Risdiplam: Infants aged between 28 days (1 month) of life and 210 days (7 months) received risdiplam orally or by bolus via naso-gastric or gastrostomy tube.
Arm/Group | Exploratory Part 1 - Risdiplam
Number analyzed (Participants) | 18
mg/kg | 0.2

2. Primary Outcome: Part 2: Percentage of Infants Who Are Sitting Without Support for at Least 5 Seconds as Assessed by Item 22 of the Gross Motor Scale of the Bayley Scales of Infant and Toddler Development Third Edition (BSID-III) at Month 12
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Item 22 is not considered achieved if the infant sits alone for less than 5 seconds before losing balance and falling over, or if the infant uses his or her arms to prop him- or herself up. The assessment was video recorded at study sites and reviewed/scored by two independent raters. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12
Population: The intent-to-treat (ITT) population is defined as all infants enrolled in Part 2 of the study, regardless of whether they received treatment or not.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 29.3 [17.84 to 43.07]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 5% derived from natural history data; p < 0.0001, One-sided Exact Binomial Test

3. Secondary Outcome: Part 2: Percentage of Infants Who Achieve a Score of 40 or Higher in the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) at Month 12
Description: The CHOP-INTEND instrument was developed to evaluate motor function in infants with SMA from the ages of 1.4 to 37.9 months. It consists of 16 items, where each item assesses a specific motor task graded on a scale of 0 to 4, where zero is no response and 4 is a complete response. The total score ranges from 0 to 64, with higher scores consistent with better motor function. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 56.1 [42.13 to 69.38]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 17% derived from natural history data; p < 0.0001, One-sided Exact Binomial Test

4. Secondary Outcome: Part 2: Percentage of Infants Achieving an Increase of >/= 4 Points in Their CHOP-INTEND Score From Baseline at Months 8 and 12
Description: as for outcome 3
Time Frame: Month 8, Month 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 8 | 87.8 [76.05 to 95.07]
  Month 12 | 90.2 [79.05 to 96.60]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 17% derived from natural history data. Statistical analysis was only performed for Month 12 data; p < 0.0001, One-sided Exact Binomial Test

5. Secondary Outcome: Part 2: Percentage of Infants Achieving Head Control (Defined as a Score of >/= 3 for CHOP-INTEND Item 12) at Months 8, 12 and 24
Description: as for outcome 3
Time Frame: Month 8, Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 8 | 46.3 [32.87 to 60.23]
  Month 12 | 53.7 [39.77 to 67.13]
  Month 24 | 70.7 [56.93 to 82.16]

6. Secondary Outcome: Part 2: Change From Baseline in the Total Raw Score of the BSID-III Gross Motor Scale at Months 12 and 24
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). In this study the gross motor scale was assessed in a modified way compared with the standard administration. A total raw score was calculated by summing the item scores to give a maximum possible score of 72.
Time Frame: Baseline, Month 12, Month 24
Population: The intent-to-treat (ITT) population is defined as all infants enrolled in Part 2 of the study, regardless of whether they received treatment or not. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Scores on a Scale
  Baseline | 1.85 (1.61)
  Change from Baseline at Month 12: number analyzed (Participants) | 38
  Change from Baseline at Month 12 | 7.21 (5.71)
  Change from Baseline at Month 24: number analyzed (Participants) | 38
  Change from Baseline at Month 24 | 12.89 (6.89)

7. Secondary Outcome: Part 2: Percentage of Infants Who Achieve the Attainment Levels of a Subset of Motor Milestones Assessed in the Hammersmith Infant Neurological Examination Module 2 (HINE-2) at Month 8
Description: The HINE was designed to evaluate infants between 2 months and 24 months of age. It is a simple and standardized instrument that includes 26 items assessing different aspects of neurological examinations, such as cranial nerves, posture, movements, tone, and reflexes. In this study, Module 2 of the HINE (HINE-2) was assessed. The HINE-2 evaluates 8 developmental milestones (head control, sitting, voluntary grasp, ability to kick, rolling, crawling, standing, and walking) scored on a 3, 4, or 5-point scale, with 0 indicating inability to perform a task and a score of 2, 3, or 4 (depending on the task) indicating full milestone development. The total score is calculated by summing the item scores to give a maximum possible score of 26. This measure represents subset numbers at Month 8 for head control, ability to kick and rolling milestones only.
Time Frame: Month 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Unable to maintain head upright (Head Control) at Month 8 | 36.6
  Wobbles (Head Control) at Month 8 | 14.6
  All the time maintained upright (Head Control) at Month 8 | 39.0
  No kicking (Ability to Kick [supine]) at Month 8 | 24.4
  Kicks horizontally; legs do not lift (Ability to Kick [supine]) at Month 8 | 58.5
  Upward (vertically) (Ability to Kick [supine]) at Month 8 | 7.3
  Touches leg (Ability to Kick [supine]) at Month 8 | 0
  Touches toes (Ability to Kick [supine]) at Month 8 | 0
  No rolling (Rolling) at Month 8 | 56.1
  Rolling to side (Rolling) at Month 8 | 29.3
  Prone to supine (Rolling) at Month 8 | 2.4
  Supine to prone (Rolling) at Month 8 | 2.4

8. Secondary Outcome: Part 2: Percentage of Infants Who Achieve the Attainment Levels of the Motor Milestones Assessed in the Hammersmith Infant Neurological Examination Module 2 (HINE-2) at Month 12
Description: The HINE was designed to evaluate infants between 2 months and 24 months of age. It is a simple and standardized instrument that includes 26 items assessing different aspects of neurological examinations, such as cranial nerves, posture, movements, tone, and reflexes. In this study, Module 2 of the HINE (HINE-2) was assessed. The HINE-2 evaluates 8 developmental milestones (head control, sitting, voluntary grasp, ability to kick, rolling, crawling, standing, and walking) scored on a 3, 4, or 5-point scale, with 0 indicating inability to perform a task and a score of 2, 3, or 4 (depending on the task) indicating full milestone development. The total score is calculated by summing the item scores to give a maximum possible score of 26.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Unable to maintain head upright (Head Control) at Month 12 | 17.1
  Wobbles (Head Control) at Month 12 | 31.7
  All the time maintained upright (Head Control) at Month 12 | 43.9
  Cannot sit (Sitting) at Month 12 | 31.7
  Sits with support at hips (Sitting) at Month 12 | 17.1
  Props (Sitting) at Month 12 | 19.5
  Stable sit (Sitting) at Month 12 | 14.6
  Pivots (rotates) (Sitting) at Month 12 | 9.8
  No grasp (Voluntary Grasp) at Month 12 | 2.4
  Uses whole hand (Voluntary Grasp) at Month 12 | 29.3
  Index finger and thumb but immature grasp (Voluntary Grasp) at Month 12 | 48.8
  Pincer grasp (Voluntary Grasp) at Month 12 | 12.2
  No kicking (Ability to Kick [supine]) at Month 12 | 12.2
  Kicks horizontally; legs do not lift (Ability to Kick [supine]) at Month 12 | 58.5
  Upward (vertically) (Ability to Kick [supine]) at Month 12 | 7.3
  Touches leg (Ability to Kick [supine]) at Month 12 | 4.9
  Touches toes (Ability to Kick [supine]) at Month 12 | 9.8
  No rolling (Rolling) at Month 12 | 36.6
  Rolling to side (Rolling) at Month 12 | 31.7
  Prone to supine (Rolling) at Month 12 | 14.6
  Supine to prone (Rolling) at Month 12 | 9.8
  Does not lift head (Crawling) at Month 12 | 85.4
  On elbow (Crawling) at Month 12 | 2.4
  On outstretched hand (Crawling) at Month 12 | 2.4
  Crawling flat on abdomen (Crawling) at Month 12 | 0
  Crawling on hands and knees (Crawling) at Month 12 | 0
  Cannot test (Crawling) at Month 12 | 2.4
  Does not support weight (Standing) at Month 12 | 61.0
  Supports weight (Standing) at Month 12 | 17.1
  Stands with support (Standing) at Month 12 | 4.9
  Stands unaided (Standing) at Month 12 | 0
  Cannot test (Standing) at Month 12 | 4.9
  Not done (Standing) at Month 12 | 4.9
  Bouncing (Walking) at Month 12 | 2.4
  Cruising (walks holding on) (Walking) at Month 12 | 0
  Walking independently (Walking) at Month 12 | 0
  Cannot test (Walking) at Month 12 | 82.9
  Not Done (Walking) at Month 12 | 7.3

9. Secondary Outcome: Part 2: Percentage of Infants Who Achieve the Attainment Levels of the Motor Milestones Assessed in the Hammersmith Infant Neurological Examination Module 2 (HINE-2) at Month 24
Description: as for outcome 8
Time Frame: Month 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Unable to maintain head upright (Head Control) at Month 24 | 7.3
  Wobbles (Head Control) at Month 24 | 19.5
  All the time maintained upright (Head Control) at Month 24 | 63.4
  Not done (Head Control) at Month 24 | 2.4
  Cannot sit (Sitting) at Month 24 | 19.5
  Sits with support at hips (Sitting) at Month 24 | 7.3
  Props (Sitting) at Month 24 | 9.8
  Stable sit (Sitting) at Month 24 | 24.4
  Pivots (rotates) (Sitting) at Month 24 | 29.3
  Not done (Sitting) at Month 24 | 2.4
  No grasp (Voluntary Grasp) at Month 24 | 2.4
  Uses whole hand (Voluntary Grasp) at Month 24 | 4.9
  Index finger and thumb but immature grasp (Voluntary Grasp) at Month 24 | 39.0
  Pincer grasp (Voluntary Grasp) at Month 24 | 41.5
  Not done (Voluntary Grasp) at Month 24 | 4.9
  No kicking (Ability to Kick [supine]) at Month 24 | 7.3
  Kicks horizontally; legs do not lift (Ability to Kick [supine]) at Month 24 | 31.7
  Upward (vertically) (Ability to Kick [supine]) at Month 24 | 9.8
  Touches leg (Ability to Kick [supine]) at Month 24 | 9.8
  Touches toes (Ability to Kick [supine]) at Month 24 | 31.7
  Not Done (Ability to Kick [supine]) at Month 24 | 2.4
  No rolling (Rolling) at Month 24 | 9.8
  Rolling to side (Rolling) at Month 24 | 29.3
  Prone to supine (Rolling) at Month 24 | 7.3
  Supine to prone (Rolling) at Month 24 | 43.9
  Not Done (Rolling) at Month 24 | 2.4
  Does not lift head (Crawling) at Month 24 | 75.6
  On elbow (Crawling) at Month 24 | 7.3
  On outstretched hand (Crawling) at Month 24 | 2.4
  Crawling flat on abdomen (Crawling) at Month 24 | 0
  Crawling on hands and knees (Crawling) at Month 24 | 4.9
  Not done (Crawling) at Month 24 | 2.4
  Does not support weight (Standing) at Month 24 | 63.4
  Supports weight (Standing) at Month 24 | 12.2
  Stands with support (Standing) at Month 24 | 14.6
  Stands unaided (Standing) at Month 24 | 0
  Not done (Standing) at Month 24 | 2.4
  Bouncing (Walking) at Month 24 | 2.4
  Cruising (walks holding on) (Walking) at Month 24 | 2.4
  Walking independently (Walking) at Month 24 | 0
  Cannot test (Walking) at Month 24 | 75.6
  Not Done (Walking) at Month 24 | 12.2

10. Secondary Outcome: Part 2: Percentage of Motor Milestone Responders as Assessed by HINE-2 at Months 12 and 24
Description: The HINE-2 evaluates 8 developmental milestones scored on a 3, 4, or 5-point scale, with 0 indicating inability to perform a task and a score of 2, 3, or 4 (depending on the task) indicating full milestone development. The total score is calculated by summing the item scores to give a maximum possible score of 26. For the motor milestone responder definition, an improvement in a motor milestone is defined as at least a 2-point increase in ability to kick (or maximal score) or a 1-point increase in head control, rolling, sitting, crawling, standing, or walking. Worsening is similarly defined as a 2-point decrease in ability to kick (or lowest score) or a 1-point decrease in head control, rolling, sitting, crawling, standing, or walking. Voluntary grasp is excluded from the definition. An infant is classified as a responder if more motor milestones show improvement than show worsening. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 78.0 [64.82 to 88.04]
  Month 24 | 85.4 [73.15 to 93.43]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 12% derived from natural history data. Statistical analysis was only performed for Month 12 data; p < 0.0001, One-sided Exact Binomial Test

11. Secondary Outcome: Part 2: Highest Motor Milestone Achieved of Six Specified Milestones Assessed in the BSID-III Gross Motor Scale by Months 12 and 24
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). This specific measure included 6 milestones: Item 9 'Controls head while upright for 15 seconds', Item 14 'Rolls from side to back', Item 22 'Sits without support for 5 seconds', Item 30 'Crawls on stomach', Item 40 'Stands alone' and Item 42 'Walks alone'. Reported here is the percentage of participants for whom the reported item was the highest item achieved out of these six items by Months 12 and 24.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Item 9: Controls Head While Upright for 15 sec at Month 12 | 0
  Item 14: Rolls from Side to Back at Month 12 | 56.1
  Item 22: Sits Without Support for 5 sec at Month 12 | 29.3
  Item 30: Crawls on Stomach at Month 12 | 0
  Item 40: Stands Alone at Month 12 | 0
  Item 42: Walks Alone at Month 12 | 0
  Item 9: Controls Head While Upright for 15 sec at Month 24 | 0
  Item 14: Rolls from Side to Back at Month 24 | 29.3
  Item 22: Sits Without Support for 5 sec at Month 24 | 61.0
  Item 30: Crawls on Stomach at Month 24 | 0
  Item 40: Stands Alone at Month 24 | 0
  Item 42: Walks Alone at Month 24 | 0

12. Secondary Outcome: Part 2: Percentage of Infants Who Are Sitting Without Support for at Least 5 Seconds as Assessed by Item 22 of the BSID-III Gross Motor Scale at Month 24
Description: as for outcome 2
Time Frame: Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 61.0 [46.94 to 73.77]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 5% derived from natural history data; p < 0.0001, One-sided Exact Binomial Test

13. Secondary Outcome: Part 2: Percentage of Infants Who Are Sitting Without Support for at Least 30 Seconds as Assessed by Item 26 of the BSID-III Gross Motor Scale at Month 24
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Item 26 is not considered achieved if the infant sits alone for less than 30 seconds before losing balance and falling over, or if the infant uses his or her arms to prop him- or herself up. The assessment was video recorded at study sites and reviewed/scored by two independent raters. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 43.9 [30.62 to 57.87]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 5% derived from natural history data; p < 0.0001, One-sided Exact Binomial Test

14. Secondary Outcome: Part 2: Percentage of Infants Who Are Standing Alone as Assessed by Item 40 of the BSID-III Gross Motor Scale at Month 24
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Reported here is the percentage of participants who achieved item 40 'Stands alone' at Month 24. The assessment was video recorded at study sites and reviewed/scored by two independent raters. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 0 [0.00 to 7.05]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 5% derived from natural history data; p = 1.0000, One-sided Exact Binomial Test

15. Secondary Outcome: Part 2: Percentage of Infants Who Are Walking Alone as Assessed by Item 42 of the BSID-III Gross Motor Scale at Month 24
Description: The BSID-III is a standardized assessment commonly used to evaluate development across five domains in infants and young children aged between 1 and 42 months. The gross motor subscale of the BSID-III is evaluated based on the linear and hierarchical obtainment of motor skills, as seen in typically developing children. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Reported here is the percentage of participants who achieved item 42 'Walks alone' at Month 24. The assessment was video recorded at study sites and reviewed/scored by two independent raters. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 0 [0.00 to 7.05]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 5% derived from natural history data; p = 1.0000, One-sided Exact Binomial Test

16. Secondary Outcome: Part 2: Time to Death
Description: The median time to event was estimated using Kaplan-Meier methodology. 90% CI was estimated using the method of Brookmeyer and Crowley.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Months | NA [NA to NA] — The median time to death was not estimable as few participants had an event.

17. Secondary Outcome: Part 2: Time to Death or Permanent Ventilation
Description: Permanent ventilation is defined as >/=16 hours of non-invasive ventilation per day or intubation for >21 consecutive days in the absence of, or following the resolution of, an acute reversible event; or tracheostomy. Permanent ventilation events were reviewed and confirmed by an independent adjudication committee. The median time to event was estimated using Kaplan-Meier methodology. 90% CI was estimated using the method of Brookmeyer and Crowley.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Months | NA [NA to NA] — The median time to death or permanent ventilation was not estimable as few participants had an event.

18. Secondary Outcome: Part 2: Time to Permanent Ventilation
Description: as for outcome 17
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Months | NA [NA to NA] — The median time to permanent ventilation was not estimable as few participants had an event.

19. Secondary Outcome: Part 2: Percentage of Infants Who Are Alive Without Permanent Ventilation at Months 12 and 24
Description: Permanent ventilation is defined as >/=16 hours of non-invasive ventilation per day or intubation for >21 consecutive days in the absence of, or following the resolution of, an acute reversible event; or tracheostomy. Permanent ventilation events were reviewed and confirmed by an independent adjudication committee. Kaplan-Meier methodology was used to estimate the percentages. 90% CI was computed using the complementary log-log transformation.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 85.37 [73.35 to 92.24]
  Month 24 | 82.93 [70.54 to 90.44]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 42% derived from natural history data. Statistical analysis was only performed for Month 12 data; p < 0.0001, One-sided Z-test

20. Secondary Outcome: Part 2: Percentage of Infants Who Are Alive at Months 12 and 24
Description: Kaplan-Meier methodology was used to estimate the percentages. 90% CI was computed using the complementary log-log transformation.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 92.68 [82.16 to 97.10]
  Month 24 | 92.68 [82.16 to 97.10]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 60% derived from natural history data. Statistical analysis was only performed for Month 12 data; p = 0.0005, One-sided Z-test

21. Secondary Outcome: Part 2: Percentage of Infants Who Are Without Permanent Ventilation at Months 12 and 24
Description: as for outcome 19
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 92.29 [81.24 to 96.95]
  Month 24 | 89.65 [77.96 to 95.32]
Statistical Analysis 1: Comparison: Confirmatory Part 2 - Risdiplam; Test type: Superiority — Result compared to a performance criterion of 89% derived from natural history data. Statistical analysis was only performed for Month 12 data; p = 0.2595, One-sided Z-test

22. Secondary Outcome: Part 2: Percentage of Infants Who Achieve a Reduction of At Least 30 Degrees in Phase Angle From Baseline, as Measured by Respiratory Plethysmography (RP) at Month 12
Description: RP measures the degree of synchrony between abdominal and thoracic cage-driven breathing. The weakness of intercostal muscles leads to asynchrony of the thorax with the diaphragm, resulting in inefficient and paradoxical breathing patterns. The degree of synchrony between the movement of the chest wall and abdomen during the respiratory cycle can be expressed as the phase angle between the two compartments and measured by placing two RP bands around the thorax and abdomen. In paradoxical breathing, the phase angle is reversed compared with the normal ventilation cycle. A phase angle of 0° indicates perfect in-phase movement, while a value of 180° indicates completely out-of-phase movement between the two compartments. In this measure, 8 or more valid breaths were used to determine the phase angle at each visit; the calculation was not performed if fewer than 8 valid breaths had been measured. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants | 34.1 [21.96 to 48.13]

23. Secondary Outcome: Part 2: Percentage of Infants Not Requiring Respiratory Support (Invasive or Non-Invasive) at Months 12 and 24
Description: 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 24.4 [13.87 to 37.85]
  Month 24 | 19.5 [10.10 to 32.46]

24. Secondary Outcome: Part 2: Percentage of Infants Able to Feed Orally at Months 12 and 24
Description: Able to feed orally includes participants fed orally and participants fed via a combination of oral and tube feeding. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Percentage of Participants
  Month 12 | 82.9 [70.31 to 91.70]
  Month 24 | 85.4 [73.15 to 93.43]

25. Secondary Outcome: Part 1 and Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From first dose up to 30 days after last dose of risdiplam (up to 60 months)
Population: All infants who received at least one dose of study medication (risdiplam) were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Exploratory Part 1 - Cohort 1 | Exploratory Part 1 - Cohort 2 | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 4 | 17 | 41
Participants
  With at least one AE | 4 | 17 | 41
  With at least one SAE | 4 | 13 | 34

26. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs Leading to Treatment Discontinuation
Description: as for outcome 25
Time Frame: From first dose up to 30 days after last dose of risdiplam (up to 60 months)
Population: All infants who received at least one dose of study medication (risdiplam) were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Participants
  Due to AE | 0
  Due to SAE | 0

27. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs Leading to Treatment Modification/Interruption
Description: as for outcome 25
Time Frame: From first dose up to 30 days after last dose of risdiplam (up to 60 months)
Population: All infants who received at least one dose of study medication (risdiplam) were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
Participants
  Due to AE | 4
  Due to SAE | 2

28. Secondary Outcome: Part 2: Anthropometric Examination of Weight Measured in Kilograms
Description: Anthropometric examination included weight, height, head circumference and chest circumference.
Time Frame: Month 12, Month 24
Population: All infants who received at least one dose of study medication (risdiplam) were included in the safety population. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 38
kilogram (kg)
  Month 12 | 9.59 (1.40)
  Month 24: number analyzed (Participants) | 36
  Month 24 | 11.28 (1.91)

29. Secondary Outcome: Part 2: Anthropometric Examination of Height, Head Circumference and Chest Circumference Measured in Centimeters
Description: Anthropometric examination included weight, height, head circumference and chest circumference.
Time Frame: Month 12, Month 24
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 38
centimeter (cm)
  Height at Month 12 | 80.47 (4.00)
  Height at Month 24: number analyzed (Participants) | 36
  Height at Month 24 | 89.13 (5.12)
  Head Circumference at Month 12 | 47.09 (1.72)
  Head Circumference at Month 24: number analyzed (Participants) | 35
  Head Circumference at Month 24 | 49.28 (2.13)
  Chest Circumference at Month 12 | 45.77 (2.31)
  Chest Circumference at Month 24: number analyzed (Participants) | 34
  Chest Circumference at Month 24 | 48.35 (3.10)

30. Secondary Outcome: Part 2: Maximum Plasma Concentration (Cmax) of Risdiplam
Description: Reported here is the maximum observed concentration throughout the observation period.
Time Frame: Day 1: 2, 4, 6, 24 hours post dose; Days 14, 119, 245, 364, 427, 490, 609, 728: predose ; Days 28, 56, 182, 301, 546, 672: predose, 2, 4, 6 hours post dose
Population: All participants with at least one time point with a risdiplam concentration measurement were included in the PK analysis data set.
Measure: Median (Full Range); unit: nanograms/milliliter (ng/mL)
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 41
nanograms/milliliter (ng/mL) | 195 [67.7 to 296]

31. Secondary Outcome: Part 2: Area Under the Curve (AUC) From 0 to 24 Hours of Risdiplam at Year 5 Visit
Description: The AUC was derived by modelling & simulation via the population pharmacokinetics (PPK) method based on the Year 5 pre-dose concentration measurement only. Hence, no other timepoints have been reported.
Time Frame: Year 5 visit: pre-dose
Population: All participants with at least one time point with a risdiplam concentration measurement were included in the PK analysis data set. Only participants for whom data were collected are included in the analysis.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 35
ng*h/mL | 2560 [1820 to 3670]

32. Secondary Outcome: Part 2: Concentration at the End of a Dosing Interval (Ctrough) of Risdiplam at Year 5
Description: Ctrough at Year 5 was the last predose sample collected from each participant who had at least 1400 days of risdiplam treatment duration.
Time Frame: Predose at Year 5
Population: as for outcome 31
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 33
ng/mL | 63.1 [15.1 to 134]

33. Secondary Outcome: Part 2: Median Fold Change From Baseline in Survival of Motor Neuron (SMN) Protein Levels in Blood
Time Frame: Days 1, 28, 119, 245, 364, 609, 728, 819 and 1820
Population: All participants with at least one time point with a protein measurement were included in the pharmacodynamic (PD) analysis data set. Only participants for whom data were collected are included in the analysis.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Confirmatory Part 2 - Risdiplam
Number analyzed (Participants) | 40
ng/mL
  Day 1 | 1.00 [1.00 to 1.00]
  Day 28: number analyzed (Participants) | 39
  Day 28 | 2.13 [0.75 to 4.66]
  Day 119: number analyzed (Participants) | 34
  Day 119 | 2.21 [0.60 to 6.33]
  Day 245: number analyzed (Participants) | 35
  Day 245 | 2.26 [0.58 to 4.54]
  Day 364: number analyzed (Participants) | 35
  Day 364 | 1.99 [0.90 to 4.06]
  Day 609: number analyzed (Participants) | 22
  Day 609 | 1.69 [1.02 to 3.67]
  Day 728: number analyzed (Participants) | 28
  Day 728 | 1.84 [0.95 to 4.25]
  Day 819: number analyzed (Participants) | 2
  Day 819 | 2.05 [1.87 to 2.23]
  Day 1820: number analyzed (Participants) | 29
  Day 1820 | 1.69 [0.72 to 4.74]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose of risdiplam (up to 60 months)
Description: All infants who received at least one dose of risdiplam were included in the safety population.
Arm/Group | Exploratory Part 1 - Cohort 1 | Exploratory Part 1 - Cohort 2 | Confirmatory Part 2 - Risdiplam
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/17 | 3/41
Serious Adverse Events (participants affected / at risk) | 4/4 | 13/17 | 34/41
Other Adverse Events (participants affected / at risk) | 3/4 | 17/17 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Part 1 - Cohort 1 (N=4) | Exploratory Part 1 - Cohort 2 (N=17) | Confirmatory Part 2 - Risdiplam (N=41)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 5 (6) | 21 (38)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Laryngeal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Part 1 - Cohort 1 (N=4) | Exploratory Part 1 - Cohort 2 (N=17) | Confirmatory Part 2 - Risdiplam (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 2 (2)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Precocious puberty (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Macular cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 12 (21)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 8 (10) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (3)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 5 (7) | 3 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (12) | 6 (13)
Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (28) | 14 (43) | 23 (66)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 9 (14)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 9 (9)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Ear infection (Infections and infestations) | 1 (1) | 3 (5) | 2 (3)
Ear, nose and throat infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (4) | 6 (8)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (14) | 11 (22)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 6 (6)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 7 (8)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 5 (8) | 7 (10)
Rotavirus infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (7) | 13 (29) | 24 (71)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 8 (9)
Varicella post vaccine (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 1 (1)
Central sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (14) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 2 (3)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02913482/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02913482/SAP_001.pdf